CLINICAL TRIAL: NCT06180551
Title: Homburg Renal Evaluation Study on the Clinical Utility of Early AKI Diagnosis
Acronym: RESCUE-AKI
Status: Recruiting | Type: Observational
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Sponsor
Other Study IDs: IMED IV-001
Record Dates: First submitted 2023-12-12; First posted 2023-12-22 (Actual); Last update posted 2023-12-22 (Actual); Status verified 2023-12

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Plasma and urine samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DKK-3 — DKK-3-Urine measurement

SUMMARY:
Critically ill patients are at risk of developing a sudden decrease of kidney function which may be detected by a decrease in urine output or is diagnosed on the basis of blood tests for substances normally eliminated by the kidney, primarily creatinine.

Because it takes about 24 hours for the creatinine level to rise, even if both kidneys have ceased to function, better markers are needed.

This trial is investigating if the marker urinary dickkopf-3 (uDKK3) allows an early prediction of a sudden decrease of kidney function.

DETAILED DESCRIPTION:
Urinary dickkopf-3 (uDKK3), a stress-induced renal tubular epithelium-derived glycoprotein, has been identified as a biomarker predicting persistent kidney dysfunction.

In this prospective observational trial in patients at high risk of developing acute kidney injury we will assess whether urinary dickkopf-3 serves as a predictor of acute kidney injury.

Patients of the intensive care units of Saarland University Hospital will be surveyed for up to two years after their admission to the intensive care unit.

The progression of the estimated Glomerular Filtration Rate and uDKK3 will be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated on the intensive care units of Saarland University Hospital.

Exclusion Criteria:

* Patients on renal replacement treatment before admission to the intensive care unit.
* Patients with chronic kidney disease stage CKD G3b or below.
* Known kidney disease.
* Kidney transplantation.
* Intoxications leading to dialysis treatment.
* Participation in other clinical trials.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients on intensive care units of the Saarland University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Urinary dickkopf-3 | Throughout observational period, defined as timeframe from admission to intensive care unit up to two years after.
  Urinary dickkopf-3
Estimated Glomerula Filtration Rate | Throughout observational period, defined as timeframe from admission to intensive care unit up to two years after.
  Estimated Glomerula Filtration Rate by CKD-EPI-formula.

SECONDARY OUTCOMES:
Mortality | Throughout observational period, defined as timeframe from admission to intensive care unit up to two years after.
  Number of patients who die during the observational period.
End Stage Renal Disease | Throughout observational period, defined as timeframe from admission to intensive care unit up to two years after.
  Number of patients with initiation of chronic kidney replacement therapy (maintenance dialysis or kidney transplantation).
Length of renal replacement therapy | During the ICU stay.
  Length of time patients receive renal replacement therapy for chronic kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Neuhaus, MD, Principal Investigator — Universität des Saarlandes
Locations (1):
- Universitätsklinikum des Saarlandes, Homburg, Saarland, Germany

IPD SHARING:
Plan to Share IPD: No